CLINICAL TRIAL: NCT02631798
Title: Mucosal Staining After Oral Administration of Food Grade Dyes in Subjects Undergoing Outpatients Colonoscopy
Brief Title: Chromocolonoscopy With Food-grade Dyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Mark Ellrichmann, Head of Interdisciplinary Endoscopy, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Microcapsule Chromo-122015
Record Dates: First submitted 2015-12-04; First posted 2015-12-16 (Estimated); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Chromoendoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dye staining (Experimental): Food grade dye mucosal staining
  Interventions: Dietary Supplement: Food grade dye mucosal staining

INTERVENTIONS:
Dietary Supplement: Food grade dye mucosal staining — mucosal staining with food grade dye

SUMMARY:
Previous with methylene blue suggested that oral administration may be superior to conventional spray catheters. The main advantages claimed were better staining due to longer exposure to the dye, more uniform staining due to normal position of the intestines (during conventional chromocolonoscopy, patients are lying on one side), and a quicker and more comfortable procedure for the patients and endoscopy personnel.

Using food-grade dyes would enable higher dye loads and lower systemic side effects.

Food grade dyes will be administered orally during preparation with KleanPrep (total amount of 4 liters) in patients undergoing screening colonoscopy.

On day 1 patients will drink 3 l of the preparation solution, the last liter together with the last dose of dye will be administered 5 hours before scheduled colonoscopy.

Primary endpoints:

* quality of mucosal staining of colon (assessed by questionnaire)

Secondary endpoints:

* adenoma detection rate
* adverse events
* time of colonoscopy

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and post-menopausal females aged 18 to 75 y and scheduled for screening colonoscopy
* body weight ≥60 kg
* good health based on medical history, physical examination, a 12-lead electrocardiogram (ECG) and routine haematology and blood chemistry tests
* ability to understand and comply with the protocol
* written informed consent

Exclusion Criteria:

* standard criteria for bioavailability estimation of new drugs, namely (i) intake of any medication, (ii) a history of drug, caffeine (>5 cups coffee/tea/day) or tobacco (≥10 cigarettes/day) abuse, (iii) history of alcohol consumption in excess of two drinks per day in males and one drink per day in females
* known or suspected hypersensitivity to food colourants,
* GI obstruction or perforation
* serious cardiovascular, renal or hepatic disease
* prolonged prothrombin time, elevated INR (international normalized ration)
* elevated serum creatinine
* any other severe underlying medical condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Quality of mucosal staining | Day of scheduled endoscopy
  Assessment of mucosal staining by questionnaire

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | Day of scheduled endoscopy and within 3 days after colonoscopy
Number of patients with detected adenomas | Day of scheduled endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ellrichmann, MD, Principal Investigator — University Hospital Schleswig-Holstein; Stefan Schreiber, Prof., Study Director — University Hospital Schleswig-Holstein
Locations (1):
- University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Schleswig-Holstein, Germany